CLINICAL TRIAL: NCT03968484
Title: Platelet Transfusion in Sepsis Trial (PlaTiSep)
Brief Title: Platelet Transfusion in Sepsis Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 trials gained priority
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PlaTiSep
Record Dates: First submitted 2019-05-29; First posted 2019-05-30 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2019-05

CONDITIONS: Sepsis; Thrombocytopenia
MeSH Terms: conditions — Sepsis; Thrombocytopenia | interventions — Platelet Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- <50.000/µl (Experimental): Transfusion of platelets starting with a platelet count <50.000/µl
  Interventions: Biological: platelet transfusion
- <20.000/µl (Experimental): Transfusion of platelets starting with a platelet count <20.000/µl
  Interventions: Biological: platelet transfusion

INTERVENTIONS:
Biological: platelet transfusion — Transfusion of platelets

SUMMARY:
Platelets are important mediators of an inflammatory response and a key component of the innate immune system to defend the human body against invading pathogens. However, little evidence exists regarding the number of platelets that should be used als transfusion threshold in septic patients. In this trial platelet transfusion will be performed with either <50000/µl or <20000/µl as a trigger.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis defined as alteration of SOFA score (Sepsis-related organ failure assessment score) >2 points (Sepsis-3 definition)
* platelet count <50.000/µl

Exclusion Criteria:

* Age less than 18 years
* patients with immune thrombocytopenia
* major bleeding in the last 72 hours or ongoing major bleeding
* patient, surrogate or physician not committed to full intensive care support
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival in 90 day follow-up period | 90 days
  overall survival at 90 days

SECONDARY OUTCOMES:
all cause mortality at 6 months | 6 months
  overall survival at 6 months
resolution of shock | 5 days
  time to normalization of lactate levels and end of vasopressor therapy
ICU length of stay | 28 days
  length of stay on ICU ward
duration of mechanical ventilation support | 28 days
  time to extubation
renal replacement therapy | 28 days
  frequency and duration of renal replacement therapy
bleeding events | 28 days
  bleeding events requiring transfusion during ICU stay
SOFA score | 28 days
  Sepsis-related organ failure assessment score
discharge location | 90 days
  discharge to home, ward, rehabilitation unit, nursing home

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenberger, Prof., Principal Investigator — University Hospital Tübingen

IPD SHARING:
Plan to Share IPD: No